CLINICAL TRIAL: NCT06323577
Title: Comparison of Functional Outcomes in Restricted Kinematic Alignment and Mechanical Alignment in Robotic Assisted Simultaneous Bilateral Total Knee Arthroplasty. A Randomized Controlled Trial
Brief Title: Comparing Efficacy Between Restricted Kinematic Alignment vs Mechanical Alignment in Bilateral TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Yot Tanariyakul, Principle investigator, Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TUH rKA vs MA TKA
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee; TKA
Keywords: restrict kinematic alignment; mechanical alignment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted kinematic alignment (Experimental)
  Interventions: Procedure: Restricted kinematic alignment
- Mechanical alignment (Active Comparator)
  Interventions: Procedure: Mechanical alignment

INTERVENTIONS:
Procedure: Restricted kinematic alignment — TKA using restricted kinematic alignment under robotic assisted surgery (MAKO).
  Arms: Restricted kinematic alignment
Procedure: Mechanical alignment — TKA using mechanical alignment under robotic assisted surgery (MAKO).
  Arms: Mechanical alignment

SUMMARY:
The goal of this RCT is to investigate efficacy between restricted kinematic alignment and mechanical alignment TKA in simultaneous bilateral TKA patients.

The main question[s] it aims to answer are:

* Does rKA have better functional outcomes than MA in simultaneous bilateral TKA patients?
* Does rKA have lower pain score than MA in simultaneous bilateral TKA patients? Participants will undergo simultaneous bilateral TKA and randomized one side will use rKA and the other side will use MA.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years
* Diagnosis bilateral primary osteoarthritis of knee joint and undergo simultaneous bilateral total knee arthroplasty
* ASA classification I-II

Exclusion Criteria:

* Valgus deformity
* BMI > 40kg/m2
* History of previous knee surgery
* Active infection of the knee joint

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-14 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Forgotten joint score | 6 weeks, 3months, 6 months, 1 year and 2 years after surgery
  Point 0-100 (0 mean worst, 100 mean best)

SECONDARY OUTCOMES:
Modified WOMAC score | 6 weeks, 3months, 6 months, 1 year and 2 years after surgery
  Point 0-96 (0 mean best, 100 mean worst)
Range of motion | 6 weeks, 3months, 6 months, 1 year and 2 years after surgery
  Using long arm goniometer (degrees)
Pain score | every 6 hours for 2 days after surgery then once a day for 2 weeks after surgery then once a week until 3 months after surgery
  Using visual analog scale (0-10, 0 mean best, 10 mean worst)
Hip knee ankle angle | 6 weeks, 3months, 6 months, 1 year and 2 years after surgery
  Evaluate by long radiograph (degrees)
Complications | Until 2 years after surgery
  For example periprosthetic fracture, infection or aspetic loosening
Incidence of soft tissue releasing | During surgery
  Record soft tissue releasing intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elbuluk AM, Jerabek SA, Suhardi VJ, Sculco PK, Ast MP, Vigdorchik JM. Head-to-Head Comparison of Kinematic Alignment Versus Mechanical Alignment for Total Knee Arthroplasty. J Arthroplasty. 2022 Aug;37(8S):S849-S851. doi: 10.1016/j.arth.2022.01.052. Epub 2022 Jan 31. PMID 35093548
- [Background] McEwen PJ, Dlaska CE, Jovanovic IA, Doma K, Brandon BJ. Computer-Assisted Kinematic and Mechanical Axis Total Knee Arthroplasty: A Prospective Randomized Controlled Trial of Bilateral Simultaneous Surgery. J Arthroplasty. 2020 Feb;35(2):443-450. doi: 10.1016/j.arth.2019.08.064. Epub 2019 Sep 5. PMID 31591010
- [Background] Van Essen J, Stevens J, Dowsey MM, Choong PF, Babazadeh S. Kinematic alignment results in clinically similar outcomes to mechanical alignment: Systematic review and meta-analysis. Knee. 2023 Jan;40:24-41. doi: 10.1016/j.knee.2022.11.001. Epub 2022 Nov 17. PMID 36403396